CLINICAL TRIAL: NCT01299519
Title: Progressive Weight Loss and Metabolic Health
Acronym: PWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201012904
Record Dates: First submitted 2011-02-10; First posted 2011-02-18 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Insulin Resistance; Obesity
Keywords: obesity; weight loss; insulin resistance
MeSH Terms: conditions — Insulin Resistance; Obesity; Weight Loss | interventions — Body Weight Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Loss (Experimental): Half of the subjects in the weight loss arm will lose 5% of their weight through a low-calorie diet, and half will also lose 10% and 15% body weight.
  Interventions: Behavioral: Weight Loss
- Weight Maintenance (Active Comparator): Subjects in the weight maintenance arm will maintain a steady body weight (plus or minus 2% of initial body weight) for six months.
  Interventions: Behavioral: Weight Maintenance

INTERVENTIONS:
Behavioral: Weight Maintenance — Subjects in the weight maintenance arm will maintain a steady body weight (plus or minus 2% of initial body weight) for six months.
  Arms: Weight Maintenance
Behavioral: Weight Loss — Half of the subjects in the weight loss arm will lose 5% of their weight through a low-calorie diet, and half will also lose 10% and 15% body weight.
  Arms: Weight Loss

SUMMARY:
This study will evaluate the potential beneficial cardiometabolic effect of moderate (5%) weight loss and progressive (5%, 10%, and 15%) weight loss in obese adults without diabetes. Participants will be randomly assigned to one of 2 groups. Group 1: supervised weight loss group (low-calorie diet). Group 2: supervised weight maintenance group (normal diet). Of those assigned to group 1, half of the participants will lose 5% of their body weight and the other half will lose 5%, 10%, and 15% of their weight over time under the guidance of a dietitian. Research testing will be repeated at each time point (5%, 10%, and 15% weight loss). In group 2, research testing will be repeated after six months.

ELIGIBILITY:
Inclusion Criteria:

* Obese: Body Mass Index from 30 to 45
* Insulin Resistant: HOMA-IR score greater than or equal to 2

Exclusion Criteria:

* diabetes
* smoking
* pregnancy
* breastfeeding
* heart failure
* history of liver disease including hepatitis
* alcoholism
* exercise more than 2 hours per week

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-02; Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | baseline through weight loss (approximately one year)
  In the weight-loss arm we will measure insulin sensitivity at baseline, after 5% weight loss, after 10% weight loss and again after 15% weight loss. Each weight loss phase will last an average of four months for a total of approximately one year. In the weight maintenance arm we will measure insulin sensitivity at baseline and after six months.
intra-hepatic triglyceride | baseline through weight loss (approximately one year)
  In the weight-loss arm we will measure intra-hepatic triglyceride at baseline, after 5% weight loss, after 10% weight loss and again after 15% weight loss. Each weight loss phase will last an average of four months for a total of approximately one year. In the weight maintenance arm we will measure intra-hepatic triglyceride at baseline and after six months.

SECONDARY OUTCOMES:
total cholesterol | baseline through weight loss (approximately one year)
  In the weight-loss arm we will measure total cholesterol at baseline, after 5% weight loss, after 10% weight loss and again after 15% weight loss. Each weight loss phase will last an average of four months for a total of approximately one year. In the weight maintenance arm we will measure total cholesterol at baseline and after six months.
systolic blood pressure | baseline through weight loss (approximately one year)
  In the weight-loss arm we will measure systolic blood pressure at baseline, after 5% weight loss, after 10% weight loss and again after 15% weight loss. Each weight loss phase will last an average of four months for a total of approximately one year. In the weight maintenance arm we will measure systolic blood pressure at baseline and after six months.
Cell proliferation (growth) rates in the colon - optional procedure | baseline through weight loss (approximately four months to one year)
  Colon cell proliferation rates will be determined using stable isotope labelled tracer methods in conjunction with sigmoid colon biopsy samples. In the weight-loss arm we will measure colonocyte proliferation rate at baseline, and once again after weight loss (either 5% weight loss, or 10% weight loss, or 15% weight loss; i.e. only one time after weight loss). Each weight loss phase will last an average of four months for a total of approximately one year. In the weight maintenance arm we will measure colonocyte proliferation rate at baseline and after six months.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] de Jonge L, Moreira EA, Martin CK, Ravussin E; Pennington CALERIE Team. Impact of 6-month caloric restriction on autonomic nervous system activity in healthy, overweight, individuals. Obesity (Silver Spring). 2010 Feb;18(2):414-6. doi: 10.1038/oby.2009.408. Epub 2009 Nov 12. PMID 19910943
- [Background] Volkow ND, Wang GJ, Telang F, Fowler JS, Goldstein RZ, Alia-Klein N, Logan J, Wong C, Thanos PK, Ma Y, Pradhan K. Inverse association between BMI and prefrontal metabolic activity in healthy adults. Obesity (Silver Spring). 2009 Jan;17(1):60-5. doi: 10.1038/oby.2008.469. Epub 2008 Oct 23. PMID 18948965
- [Background] McLaughlin T, Abbasi F, Kim HS, Lamendola C, Schaaf P, Reaven G. Relationship between insulin resistance, weight loss, and coronary heart disease risk in healthy, obese women. Metabolism. 2001 Jul;50(7):795-800. doi: 10.1053/meta.2001.24210. PMID 11436184
- [Derived] van Vliet S, Koh HE, Patterson BW, Yoshino M, LaForest R, Gropler RJ, Klein S, Mittendorfer B. Obesity Is Associated With Increased Basal and Postprandial beta-Cell Insulin Secretion Even in the Absence of Insulin Resistance. Diabetes. 2020 Oct;69(10):2112-2119. doi: 10.2337/db20-0377. Epub 2020 Jul 10. PMID 32651241
- [Derived] Yoshino J, Patterson BW, Klein S. Adipose Tissue CTGF Expression is Associated with Adiposity and Insulin Resistance in Humans. Obesity (Silver Spring). 2019 Jun;27(6):957-962. doi: 10.1002/oby.22463. Epub 2019 Apr 19. PMID 31004409
- [Derived] Chondronikola M, Magkos F, Yoshino J, Okunade AL, Patterson BW, Muehlbauer MJ, Newgard CB, Klein S. Effect of Progressive Weight Loss on Lactate Metabolism: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 Apr;26(4):683-688. doi: 10.1002/oby.22129. Epub 2018 Feb 24. PMID 29476613